CLINICAL TRIAL: NCT01711801
Title: A Single-Center, Randomized, Investigator/Subject-Blind, Adaptive Single-Ascending Dose, Placebo-Controlled, Parallel Study to Investigate the Safety, Tolerability, Pharmacokinetics (Including the Effect of Food), and Pharmacodynamics of RO5545965 Following Oral Administration in Healthy Subjects.
Brief Title: A Study of Safety, Pharmacokinetics (Including Food Effect) And Pharmacodynamics of RO5545965 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP28373; 2012-002869-35 (EudraCT Number)
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Part 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 1: RO5545965 (Experimental)
  Interventions: Drug: RO5545965
- Part 2: Food effect (Experimental)
  Interventions: Drug: RO5545965

INTERVENTIONS:
Drug: Placebo — Single ascending dose
  Arms: Part 1: Placebo
Drug: RO5545965 — Single ascending dose
  Arms: Part 1: RO5545965
Drug: RO5545965 — Single dose, in fed and fasted state
  Arms: Part 2: Food effect

SUMMARY:
This randomized, Investigator/Subject-blind, adaptive single-ascending-dose, placebo-controlled, parallel study will evaluate the safety, tolerability, pharmacokinetics (including the effect of food), and pharmacodynamics of RO5545965 following oral administration in healthy male volunteers. In Part 1, subjects will be randomized in cohorts to receive single ascending doses of RO5545965 or placebo. In Part 2, subjects will receive 2 doses of RO5545965, in the fed or fasted state, in randomized sequence with a washout period of approximately 2 weeks between treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, 18 to 45 years of age, inclusive. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology and urinalysis
* Body mass index (BMI) 18 to 30 kg/m2 inclusive
* Male subjects (whether surgically sterilized or not) with female partners of child-bearing potential must use two forms of contraception, one of which must be a barrier method, for the duration of the study and for 77 days after the last dose

Exclusion Criteria:

* History or presence of any clinically significant disease or disorder
* Any condition or disease that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the opinion of the investigator
* History of clinically significant hypersensitivity or allergic drug reactions
* Any suspicion or history of alcohol abuse and/or consumption of other drugs of abuse
* Regular smoker (> 5 cigarettes, > 1 pipeful or > 1 cigar per day)
* Positive for hepatitis B, hepatitis C or HIV infection
* Dietary restrictions that would prohibit the consumption of standardized meals
* Participation in an investigational drug or device study within 90 days prior to screening, as calculated from the follow-up from the previous study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | up to approximately 10 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) | Pre-dose and up to 48 hours post-dose
Pharmacokinetics: Maximum plasma concentration (Cmax) | Pre-dose and up to 48 hours post-dose
Pharmacodynamics: Prolactin levels | Pre-dose and up to 10 hours post-dose
Effect of food on the pharmacokinetics of single dose RO55459965: Area under the concentration-time curve (AUC) | pre-dose and up to 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands